CLINICAL TRIAL: NCT01319929
Title: A Proof of Concept Study of the Effects of LY2828360 in the Treatment of Patients With Osteoarthritic Knee Pain.
Brief Title: A Study of LY2828360 in Patients With Osteoarthritic Knee Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 14165; I4F-EW-CCAC (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-03-18; First posted 2011-03-22 (Estimated); Results first posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis, knee pain, osteoarthritic knee pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — CB2 receptor agonist LY2828360

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2828360 then Placebo (Experimental): 80 milligrams (mg) of LY2828360 daily by mouth for 4 weeks: placebo daily by mouth for 4 weeks. There is a washout period of 3 weeks between treatments.
  Interventions: Drug: LY2828360; Drug: Placebo
- Placebo then LY2828360 (Experimental): Placebo daily by mouth for 4 weeks: LY2828360 daily by mouth for 4 weeks. There is a washout period of 3 weeks between treatments.
  Interventions: Drug: LY2828360; Drug: Placebo

INTERVENTIONS:
Drug: LY2828360 — Administered orally
Drug: Placebo — Administered orally

SUMMARY:
To investigate the safety, efficacy and pharmacokinetics of single daily oral dose of LY2828360 in male and female subjects with osteoarthritic knee pain

ELIGIBILITY:
Inclusion Criteria:

* Are male or female participants with osteoarthritis (OA), as determined by medical history and physical examination. Males and females with stable medical problems that, in the investigator's opinion, will not significantly alter the disposition of the drug, will not place the participant at increased risk by participating in the study, and will not interfere with interpretation of the data.

  1. Male participants: agree to use a reliable method of birth control during the study and for 3 months following the last dose of the investigational product
  2. Female participants: women not of child-bearing potential due to surgical sterilization (at least 6 weeks post surgical bilateral oophorectomy with or without hysterectomy or tubal ligation) confirmed by medical history, or menopause
* Body weight greater than 40 kilograms (kg) and less than 120 kilograms (kg) with a body mass index (BMI) between 19-35 kilograms per square meter (kg/m^2) inclusive
* Participant with osteoarthritic knee based on disease diagnostic criteria as presented in the Inclusion Disease Criteria, below
* Blood pressure and pulse rate in supine and standing positions, within normal reference ranges for the population and investigator clinical research unit (CRU), or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Have clinical laboratory test results within normal reference range for the population or investigator clinical research unit (CRU), or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Have venous access sufficient to allow for blood sampling
* Have agreed to maintain the same activity level throughout the course of the study

Inclusion Disease Criteria:

* Have a unilateral or bilateral osteoarthritis (OA) of the knee diagnosed according to the American College of Rheumatology (ACR) criteria. The clinical diagnosis of osteoarthritis (OA) will be confirmed by the American College of Rheumatology (ACR) clinical and radiographic criteria for classification of idiopathic osteoarthritis (OA) of the knee based upon the following criteria:

  1. Knee pain for at least 14 days per month for the 3 months before screening
  2. Osteophytes (with radiographic evidence)
  3. At least 1 of the following 3 conditions: Age greater than 50, or Morning stiffness less than 30 minutes, or Crepitus
* Have a Kellgren and Lawrence grade of I, II, III or IV
* Have a mean score of at least 4 (moderate) and less than or equal to 8 (moderate-severe) on the 24-hour average pain score (0-10) (question 1) in the participant e-diary from screening to randomization for the knee joint during walking
* Discontinued use of all analgesic medications (including over-the-counter [OTC] analgesics/Non-Steroidal Anti-Inflammatory Drug [NSAID]) at least 2 weeks prior to randomization (participants are allowed limited use of analgesic medications)

Exclusion Criteria:

* Are currently enrolled in, have completed or discontinued within the last 3 months from, a clinical trial involving an off-label investigational drug or device or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have known allergies to LY2828360, related compounds or any components of the formulation
* Have an abnormality in the 12-lead electrocardiogram (ECG) at screening that, in the opinion of the investigator, increases the risks associated with participation in the study
* Have a recent or current history of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Have current or previous (within the past year) Axis 1 diagnosis of major depressive disorder, mania, bipolar disorder, psychosis, dysthymia, generalized anxiety disorder, alcohol or eating disorders according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition Text Revision, criteria, as determined by the investigator and confirmed by the Mini-International Neuropsychiatric Interview
* Are judged by the Principal Investigator to be clinically at suicidal risk based upon clinical interview
* Have intercurrent illness or clinically significant adverse events
* Have increased risk of seizures as evidenced by a history of seizures, stroke, surgery to the cerebral cortex, or head trauma with loss of consciousness
* Have an alanine aminotransaminase (ALT) greater than 2.5 times Upper Limit of Normal (ULN) at Screening, based on reference ranges of the local laboratory. Moderate or greater hepatic impairment
* Have prior renal transplant, current renal dialysis or severe renal insufficiency, or serum creatinine laboratory value greater than 1.5 times Upper Limit of Normal, based on the reference ranges of the local laboratory
* Have clinically significant abnormal neurological examination, especially any evidence of tremor or nystagmus
* Have a history of or symptoms suggestive of sleep apnoea
* Use of any known strong inducers or inhibitors of Cytochrome P450 within 30 days prior to enrolment.
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Have a positive alcohol breath test at Screening
* Show evidence of human immunodeficiency virus infection and/or positive human HIV antibodies
* Have an active malignancy of any type or a history of malignancy (except basal cell carcinoma of the skin that has been excised prior to study start)
* Are at a high risk of infection
* Have an autoimmune disorder
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen
* Are women with a positive pregnancy test or women who are lactating or child bearing
* Use prescription and herbal medications that cannot safely be discontinued by end of screening
* Have donated blood of more than 500 milliliters (mL) within the last 3 months
* Have an average weekly alcohol intake that exceeds 21 units per week (males up to age 65) and 14 units per week (males over 65 and females), or are unwilling to refrain alcohol consumption for the duration of the study
* Are persons who have previously received the investigational product in study, have completed or withdrawn from this study or any other study investigation LY2828360
* Are taking any excluded medications (analgesic medications) and over-the- counter medications that cannot be discontinued at screening
* Show evidence or have any prior history of significant active neurological or psychiatric disease including depression

Exclusion Disease Criteria:

* Have secondary causes of arthritis of the knee including septic arthritis, inflammatory joint disease, articular fracture, major dysplasias or congenital abnormality, ochronosis, acromegaly, hemochromatosis, Wilson's disease, and primary osteochondromatosis
* Have had lower extremity surgery (including arthroscopy of the index knee) within 6 months prior to Screening or have surgery planned of the index knee at anytime
* Have had significant prior injury to the index knee within 12 months prior to Screening
* Use of lower extremity assistive devices other than a cane or knee brace (use of a 'shoe lift' is permitted). Are non-ambulatory or require the use of crutches or a walker. Use of a cane in the hand opposite the index knee is acceptable
* Have a confounding painful condition that may interfere with assessment of the index joint, that is, knee
* Have any other musculoskeletal or arthritic condition that may affect the interpretation of clinical efficacy and/or safety data or otherwise contraindicates participation in this clinical study
* Have used corticosteroid prior to baseline
* Have received hyaluronan injections into index knee within the previous 6 months prior to Treatment Phase day 3
* Have initiated or have changed to an established physiotherapy program within 2 weeks prior to Treatment Phase day 3 or during the study period An established physiotherapy program may be continued throughout the study period if unchanged in frequency and intensity
* Has had a prior synovial fluid analysis showing a White Blood Cell (WBC) greater than or equal to 2000 cubic millimeters (mm^3) that is indicative of a diagnosis other than OA
* Have started recently or changed dose regimen of any OA specific therapies (that is, nutraceutical products)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aalborg, Denmark

RESULTS

PARTICIPANT FLOW:
Groups:
- 80 mg LY2828360 First, Then Placebo: Participants received 80 milligrams (mg) of LY2828360 once daily by mouth for 4 weeks, followed by a 3-week washout period, then placebo once daily by mouth for 4 weeks.
- Placebo First, Then 80 mg LY2828360: Participants received placebo once daily by mouth for 4 weeks, followed by a 3-week washout period, then 80 mg of LY2828360 once daily by mouth for 4 weeks.
Period: First Treatment Period (4 Weeks)
Arm/Group | 80 mg LY2828360 First, Then Placebo | Placebo First, Then 80 mg LY2828360
Started | 20 | 19
Completed | 17 | 17
Not Completed | 3 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 0 | 1
Period: Washout Period (3 Weeks)
Arm/Group | 80 mg LY2828360 First, Then Placebo | Placebo First, Then 80 mg LY2828360
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0
Period: Second Treatment Period (4 Weeks)
Arm/Group | 80 mg LY2828360 First, Then Placebo | Placebo First, Then 80 mg LY2828360
Started | 17 | 17
Completed | 16 | 16
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Sponsor Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 80 mg LY2828360 First, Then Placebo | Placebo First, Then 80 mg LY2828360 | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (6.6) | 61.9 (7.1) | 63.3 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 15 | 10 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 19 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Denmark | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 4 Week Endpoint in Weekly Mean of Daily 24-Hour Average Pain Scores (APS)
Description: The weekly mean of the 24-Hour APS was calculated from participants' daily entries for 24-hour average pain rating on an 11-point scale with scores from 0 (no pain) to 10 (worst possible pain). Data were recorded twice a day at approximately the same time each day, preferably first thing in the morning and in the afternoon.
Time Frame: Baseline, 4 weeks
Population: The analysis included all randomized participants receiving at least 1 dose of the investigational product and with a baseline and at least 1 post-baseline weekly mean 24-Hour Average Pain value.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 80 mg LY2828360: Participants received 80 milligrams (mg) of LY2828360 once daily by mouth for 4 weeks.
- Placebo: Participants received placebo once daily by mouth for 4 weeks.
Arm/Group | 80 mg LY2828360 | Placebo
Number analyzed (Participants) | 34 | 34
units on a scale | -0.90 (1.03) | -1.20 (1.50)

2. Secondary Outcome: Pharmacokinetics (PK) of LY2828360: Maximal Concentration (Cmax)
Time Frame: Pre-last dose to 8 hours post-last dose (at end of each 4-week treatment period)
Population: The analysis included all randomized participants receiving at least 1 dose of LY2828360 with interpretable PK data.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | 80 mg LY2828360
Number analyzed (Participants) | 34
nanogram per milliliter (ng/mL) | 464.4 (161.0)

3. Secondary Outcome: Pharmacokinetics (PK) of LY2828360: Area Under the Concentration-Time Curve (AUC)
Description: AUC from time zero to 8 hours (AUC0-8h) is reported for this outcome measure.
Time Frame: Pre-last dose to 8 hours post-last dose (at end of each 4-week treatment period)
Population: The analysis included all randomized participants receiving at least 1 dose of LY2828360 with interpretable PK data.
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | 80 mg LY2828360
Number analyzed (Participants) | 34
nanogram*hour per milliliter (ng*h/mL) | 2803.9 (775.8)

4. Secondary Outcome: Change From Baseline to 4 Week Endpoint in Weekly Mean of Night Pain and Worst Daily Pain Scores
Description: The pain severity for night pain and worst pain was measured by an 11-point Likert scale, an ordinal scale with scores from 0 (no pain) to 10 (worst possible pain). The 11-point Likert scale was used for assessment of night pain and worst pain each day, and evaluated as weekly means. Participants were asked to complete the severity pain for worst pain twice a day (in the morning and in the afternoon). The pain severity for night pain was filled out only once in the morning.
Time Frame: Baseline, 4 weeks
Population: The analysis included all randomized participants receiving at least 1 dose of the investigational product and with a baseline night/worst pain value and at least 1 post-baseline weekly mean night/worst pain value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 80 mg LY2828360 | Placebo
Number analyzed (Participants) | 34 | 34
units on a scale
  Night Pain | -0.80 (1.08) | -1.15 (1.47)
  Worst Daily Pain | -0.85 (1.27) | -1.25 (1.62)

5. Secondary Outcome: Change From Baseline to 4 Week Endpoint in Chronic Pain Sleep Inventory (CPSI)
Description: The CPSI is a validated 5-item questionnaire in which the following factors were assessed: trouble falling asleep due to pain (CPSI1), the need for sleep medication (CPSI2), awakenings by pain during the night (CPSI3) awakenings by pain in the morning (CPSI4), and overall sleep quality (CSPI5). All CPSI items are scored using a 100-millimeter (mm) visual analog scale (VAS) (VAS; 0=never and 100=always for CPSI1 through CPSI4, and 0=very poor and 100=excellent for CPSI5).
Time Frame: Baseline, 4 weeks
Population: The analysis included all randomized participants receiving at least 1 dose of the investigational product and with a baseline and at least 1 postbaseline CPSI value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 80 mg LY2828360 | Placebo
Number analyzed (Participants) | 34 | 34
units on a scale
  CPSI1: Trouble falling asleep due to pain | -0.6 (0.9) | -0.6 (1.2)
  CPSI2: Need for sleep medication | 0.0 (0.3) | -0.1 (0.5)
  CPSI3: Awakenings by pain during the night | -0.5 (1.2) | -0.8 (1.5)
  CPSI4: Awakenings by pain in the morning | -0.4 (1.1) | -0.7 (1.2)
  CPSI5: Overall sleep quality | 0.8 (1.4) | 1.3 (1.4)

6. Secondary Outcome: Change From Baseline to 4 Week Endpoint in Pittsburgh Sleep Quality Index (PSQI)
Description: The PSQI is a self-rated questionnaire that assesses the participant's sleep habits during the last month and consists of 19 questions that cover 7 components (sleep quality, sleep onset latency, sleep duration, sleep efficiency, sleep disturbances, sleeping medication use, and daytime dysfunction). Each item has a range of 0 (no difficulty) to 3 (severe difficulty). The 7 component scores were added to yield a global score with a range of 0 (no difficulty) to 21 (severe difficulties in all areas).
Time Frame: Baseline, 4 weeks
Population: The analysis included all randomized participants receiving at least 1 dose of the investigational product and with a baseline and at least 1 postbaseline PSQI value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 80 mg LY2828360 | Placebo
Number analyzed (Participants) | 34 | 34
units on a scale | -0.9 (2.8) | -0.7 (1.5)

7. Secondary Outcome: Change From Baseline to 4 Week Endpoint in Brief Pain Inventory Severity and Interference Scores (BPI-S/BPI-I)
Description: The BPI-S and BPI-I are self-reported scales measuring severity of pain and interference on function. BPI-S consists of 4 questions assessing worst pain, least pain, average pain in the past 24 hours, and pain right now. Severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine). The BPI-I average interference is the average of 7 questions assessing interference of pain for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Average interference scores range: 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline, 4 weeks
Population: The analysis included all randomized participants receiving at least 1 dose of the investigational product and with baseline and at least 1 postbaseline BPI-S/BPI-I value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 80 mg LY2828360 | Placebo
Number analyzed (Participants) | 34 | 34
units on a scale
  BPI-S Worst Pain | -1.0 (1.7) | -1.0 (1.9)
  BPI-S Least Pain | -0.6 (1.0) | -0.8 (1.8)
  BPI-S Average Pain in the Past 24 Hours | -0.9 (1.1) | -1.1 (1.6)
  BPI-S Pain Right Now | -0.6 (1.4) | -0.8 (1.7)
  BPI-I Average Interference | -0.7 (1.2) | -0.8 (1.2)

8. Secondary Outcome: Change From Baseline to 4 Week Endpoint in Investigator Global Assessment of Changes (IGAC)
Description: The IGAC is an investigator-reported subjective evaluation using a 100 millimeter (mm) visual analog scale (VAS) to answer the following question: If you take into consideration all the various ways the knee pain influence the participant and his/her life, how do you then evaluate the participant's condition today (0=very good and 100=very bad).
Time Frame: Baseline, 4 weeks
Population: The analysis included all randomized participants receiving at least 1 dose of the investigational product and with baseline and at least 1 postbaseline IGAC value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 80 mg LY2828360 | Placebo
Number analyzed (Participants) | 34 | 34
units on a scale | -8.6 (15.6) | -8.6 (16.2)

9. Secondary Outcome: Change From Baseline to 4 Week Endpoint in Patient Global Assessment of Changes (PGAC)
Description: The PGAC is a self-reported subjective evaluation using a 100 millimeter (mm) visual analog scale (VAS) to answer the following question: If you take into consideration all the various ways the knee pain influence you and your life how do you then evaluate your condition over the last week (0=very good and 100=very bad).
Time Frame: Baseline, 4 weeks
Population: The analysis included all randomized participants who received at least 1 dose of the investigational product and with a baseline and at least 1 postbaseline PGAC value.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 80 mg LY2828360: The analysis included all randomized participants received 80 milligrams (mg) of LY2828360 once daily by mouth for 4 weeks.
Arm/Group | 80 mg LY2828360 | Placebo
Number analyzed (Participants) | 34 | 34
units on a scale | -9.6 (21.7) | -10.5 (21.3)

10. Secondary Outcome: Change From Baseline to 4 Week Endpoint in Western Ontario and MacMaster (WOMAC)
Description: WOMAC index completed by participant; consists of 24 questions, each based on 5-point Likert scale (0=none to 4=extreme). Has 3 subscales: pain, stiffness, and physical function. Pain subscale has 5 questions on pain associated with everyday tasks; subscale score ranges from 0=none to 20=extreme. Physical function subscale has 17 questions on physical function difficulties with everyday tasks; subscale score ranges from 0=none to 68=extreme. Stiffness subscale has 2 questions on stiffness associated with time of day (morning versus later in day); subscale score ranges from 0=none to 8=extreme.
Time Frame: Baseline, 4 weeks
Population: The analysis included all randomized participants receiving at least 1 dose of the investigational product and with a baseline and at least 1 postbaseline WOMAC value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 80 mg LY2828360 | Placebo
Number analyzed (Participants) | 34 | 34
units on a scale
  WOMAC: Pain | -0.9 (2.3) | -1.6 (2.5)
  WOMAC: Stiffness | -0.5 (1.4) | -0.5 (1.5)
  WOMAC: Physical Function | -3.4 (7.8) | -3.9 (7.9)

11. Secondary Outcome: Change From Baseline to 4 Week Endpoint in Pain From 40 Meter Self-Paced Walk Test
Description: The 40 meter self-paced walk test is a participant-rated subjective evaluation using a 100 millimeter (mm) visual analog scale (VAS) to assess pain after walking 40 meters. Scores range from 0 (no pain) to 100 (worst pain).
Time Frame: Baseline, 4 weeks
Population: The analysis included all randomized participants receiving at least 1 dose of the investigational product and with a baseline and at least 1 postbaseline 40 Meter Self-Paced Walk test value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 80 mg LY2828360 | Placebo
Number analyzed (Participants) | 34 | 34
units on a scale | -7.8 (18.0) | -8.4 (24.7)

12. Secondary Outcome: Change From Baseline to 4 Week Endpoint in the 11 Step Stair Climb Test
Description: The 11 step stair climb test is a participant-rated subjective evaluation using a 100 millimeter (mm) visual analog scale (VAS) to assess pain after climbing 11 stairs. Scores range from 0 (no pain) to 100 (worst pain).
Time Frame: Baseline, 4 weeks
Population: The analysis included all randomized participants receiving at least 1 dose of investigational product and with baseline and at least 1 postbaseline 11 Step Stair Climb Test value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 80 mg LY2828360 | Placebo
Number analyzed (Participants) | 34 | 34
units on a scale | -4.0 (16.0) | -9.0 (23.9)

13. Secondary Outcome: Change From Baseline to 4 Week Endpoint in DoloTest Sum Score
Description: The DoloTest® is a self-reported assessment composed of 8 visual analog scale (VAS) items ranging from 0 (none) to 100 (worst possible) for the following domains: pain, problems with light physical activities, problems with more strenuous physical activities, problems doing your job, reduced energy and strength, low spirit, reduced social life, and problems sleeping). The scale is arranged in a radar plot to provide a graphic presentation of the test result. The DoloTest® Sum Score is equal to the sum of each scored domain; scores range from 0 (none) to 800 (worst possible).
Time Frame: Baseline, 4 weeks
Population: The analysis included all randomized participants receiving at least 1 dose of investigational product and with a baseline and at least 1 postbaseline DoloTest value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 80 mg LY2828360 | Placebo
Number analyzed (Participants) | 34 | 34
units on a scale | -34.5 (90.0) | -51.5 (88.6)

14. Secondary Outcome: Number of Participants With Treatment-Emergent Suicidal Ideation and Behaviors Assessed by Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS: scale capturing occurrence, severity, and frequency of suicide-related thoughts and behaviors. Number of participants with suicidal behaviors and ideations are provided. Suicidal behavior: a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation: a "yes" answer to any one of 5 suicidal ideation questions, which includes wish to be dead, and 4 different categories of active suicidal ideation.
Time Frame: Baseline up to 15 weeks
Population: The C-SSRS analysis included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | 80 mg LY2828360 | Placebo
Number analyzed (Participants) | 37 | 36
Participants
  Treatment-Emergent Suicidal Ideation | 0 | 0
  Treatment-Emergent Suicidal Behaviors | 0 | 0

ADVERSE EVENTS:
Arm/Group | 80 mg LY2828360 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/36
Other Adverse Events (participants affected / at risk) | 14/37 | 16/36
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 80 mg LY2828360 (N=37) | Placebo (N=36)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (3)
Nausea (Gastrointestinal disorders) | 4 (5) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2)
Fatigue (General disorders) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (3)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 4 (5) | 1 (1)
Headache (Nervous system disorders) | 4 (5) | 2 (2)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days